CLINICAL TRIAL: NCT06906380
Title: A Long-term Follow-up Study of Patients Enrolled in ARD103_ARCE-CL-P-001 Phase 1/2 Study and Treated With ARD103 CAR-T Cell Therapies
Brief Title: A Long-term Follow-up Study of Patients With ARD103 CAR-T Cell Therapies
Status: Not yet recruiting | Type: Observational
Sponsor: ARCE Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARD103_ARCE-CL-P-002
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia, in Relapsed or Refractory; MDS (Myelodysplastic Syndrome)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non Interventional: All subjects with AML or MDS who are enrolled in a parent study and were exposed to ARD103 CAR-T cellular therapy will be asked to participate in this long-term follow-up (LTFU) study.
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Non Intervention, an observation LTFU study

SUMMARY:
This study will evaluate the long-term safety of ARD103 cellular therapies

DETAILED DESCRIPTION:
Participants who receive administration of ARD103 (i.e., a partial dose or a full dose) will roll into the LTFU study upon completion of the 24-month interventional study period (Study: ARD103_ARCE-CL-P-001), or after early discontinuation from the interventional study protocol. The LTFU study is a study intended to characterize long-term safety for 15 years post-ARD103 administration. Participants who complete the full 24-month interventional study period will undergo an additional 13 years of monitoring under the LTFU study. No IP will be administered during the LTFU study. The number and percentage of participants with ARD103 CAR-T cell therapy related AEs, SAEs, and AESIs will be recorded throughout the LTFU Period.

ELIGIBILITY:
Inclusion Criteria:

* The participant has R/R AML or MDS and has previously received ARD103 CAR-T cell therapies in the parent study.
* The participant is able to understand and comply with protocol-required study procedures and has provided a written informed consent document.

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise participants with R/R AML or MDS treated with ARD103. All subjects with AML or MDS who are enrolled in a parent study and were received ARD103 CAR-T infusion will be asked to participate in this long-term follow-up (LTFU) study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2040-05-30 (Estimated); Study Completion 2040-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and duration of AEs, SAEs, and AESIs related to ARD103 treatment. | 15 years
  The number and percentages of participants experiencing TEAEs will be tabulated. Serious TEAEs will be summarized and AESIs will be summarized.

SECONDARY OUTCOMES:
The long-term efficacy of ARD103 in participants with R/R AML or MDS | 15 years
  Overall survival (OS): the time from the infusion of ARD103 CAR-T in the parent study until death for any cause.
  Duration of Response (DOR): the time from the first recorded response after ARD103 infusion to the first recorded efficacy result of disease progression, relapse, or death due to any cause, whichever occurs first.
  PFS: the time from the infusion of ARD103 in the parent study to the first recorded response of disease progression, relapse, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute, Winston-Salem, North Carolina
  - MD Anderson Cancer Center, Houston, Texas